CLINICAL TRIAL: NCT02675946
Title: A Phase 1 Open-label Dose Escalation Study of CGX1321 in Subjects With Advanced Solid Tumors With Expansion in Advanced Gastrointestinal Tumors and Phase 1b Study of CGX1321 in Combination With Pembrolizumab in Subjects With Advanced Colorectal Cancer or in Combination With Encorafenib + Cetuximab in Subjects With BRAFV600E Mutated Advanced Colorectal Cancer
Brief Title: CGX1321 in Subjects With Advanced Solid Tumors and CGX1321 With Pembrolizumab or Encorafenib + Cetuximab in Subjects With Advanced GI Tumors (Keynote 596)
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Curegenix Inc. (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CGX1321-101; MK3475-596 (Other: Merck, Sharpe and Dohme Corporation)
Record Dates: First submitted 2016-01-22; First posted 2016-02-05 (Estimated); Last update posted 2022-01-26 (Actual); Status verified 2022-01

CONDITIONS: Solid Tumors; GI Cancer
Keywords: WNT inhibitor
MeSH Terms: conditions — Gastrointestinal Neoplasms | interventions — CGX1321; pembrolizumab; encorafenib; Cetuximab

STUDY DESIGN:
Intervention Model Description: Enrollment to Single Agent Dose Expansion, Roll-over Cohort, Phase 1b CGX1321-101 in combination with pembrolizumab dose expansion and Phase 1b CGX1321 in combination with encorafenib + cetuximab dose escalation and dose expansion
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm 1: CGX1321 Single Agent dose escalation and dose expansion (Experimental): Arm 1: Dose Escalation Phase: Ascending doses of CGX1321 once daily, orally, for 3 weeks (21 days) followed by a one-week (7-day) washout period in each 28-day cycle
  Dose Expansion Phase: CGX1321, at the MTD (identified in the Dose Escalation Phase), once daily, orally, for 3 weeks (21 days) followed by a one-week (7-day) washout period in each 28-day cycle.
  Interventions: Drug: CGX1321
- Arm 2: CGX1321 in combination with pembrolizumab dose escalation, dose expansion and Roll-over, (Experimental): Arm 2: Roll-over Cohort: CGX1321 at a dose identified in Phase 1b, once daily, orally, for 2 weeks (14 days) followed by a one-week (7-day) washout period in combination with pembrolizumab administered IV once every three weeks (in each 21-day cycle).
  Arm 2: Phase 1b: Ascending doses of CGX1321, once daily, orally, for 2 weeks (14 days) followed by a one-week (7-day) washout period in combination with pembrolizumab administered IV once every three weeks (in each 21-day cycle).
  Interventions: Drug: CGX1321; Drug: Pembrolizumab
- Arm 3: CGX1321 in combination with encorafenib + cetuximab, dose escalation and dose expansion (Experimental): Arm 3: Phase 1b: Ascending doses of CGX1321, once daily, orally for 3 weeks (21 days) followed by a one-week (7 day) washout period in combination with enocrafenib administered orally once daily and cetuximab administered IV once weekly
  Interventions: Drug: CGX1321; Drug: encorafenib; Drug: cetuximab

INTERVENTIONS:
Drug: CGX1321
Drug: Pembrolizumab
  Other Names: Keytruda
  Arms: Arm 2: CGX1321 in combination with pembrolizumab dose escalation, dose expansion and Roll-over,
Drug: encorafenib
  Other Names: Braftovi
  Arms: Arm 3: CGX1321 in combination with encorafenib + cetuximab, dose escalation and dose expansion
Drug: cetuximab
  Other Names: Erbitux
  Arms: Arm 3: CGX1321 in combination with encorafenib + cetuximab, dose escalation and dose expansion

SUMMARY:
This is a multicenter, open-label study conducted in two phases: Phase 1 consisting of a CGX1321 Single Agent Dose Escalation Phase in solid tumors, CGX1321 Single Agent Dose Expansion Phase in GI tumors and Roll-over Cohort of CGX1321 and pembrolizumab in subjects who have progressed on single agent CGX1321 and Phase 1b consisting of CGX1321 in combination with pembrolizumab in colorectal tumors and CGX1321 in combination with encorafenib + cetuximab in BRAFV600E mutated colorectal tumors. Both phases are to evaluate safety, pharmacokinetics, and clinical activity.

DETAILED DESCRIPTION:
The purpose of the Dose Escalation Phase is to examine the safety and determine the maximum tolerated dose of CGX1321 when administered to subjects with advanced solid tumors.

The purpose of the Dose Expansion Phase, Roll-over Cohort and Phase 1b is to continue to examine the safety and confirm the final Phase 2 dose of CGX1321 alone in subjects with advanced GI tumors (Dose Expansion Phase) and evaluate the safety and tolerability of CGX1321 in combination with pembrolizumab (Phase 1b and Roll-over Cohort) and of CGX1321 in combination with encorafenib + cetuxumab (Phase 1b)

ELIGIBILITY:
Inclusion Criteria The following criteria must be met by ALL subjects

1. Have measurable disease based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 (Phase 1) or immune-related (ir)RECIST 1.1 (Phase 1b and Roll-over Cohort). Tumor lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions
2. Minimum estimated life expectancy of 3 months
3. Age 18 years or older
4. Must have adequate organ function, including the following:

   * Absolute neutrophil count (ANC) ≥ 1.5 x109/L; platelet count ≥ 100 x 109/L; hemoglobin ≥ 9 g/dL or ≥ 5.6 mmol/L
   * International normalized ratio (INR) or prothrombin time (PT) and activated partial thromboplastin Time (aPTT) ≤ 1.5 times the upper limit of normal (ULN) unless subject is receiving anticoagulant therapy as long as PT or aPTT is within therapeutic range of intended use of anticoagulants
   * Hepatic: total bilirubin ≤ 1.5 times ULN, aspartate transaminase (AST) and/or alanine aminotransferase (ALT) ≤ 2.5 times ULN (≤ 5 times ULN if liver metastases)
   * Renal: serum creatinine ≤ 1.25 times the ULN or estimated creatinine clearance ≥ 60 mL/min (Cockcroft and Gault formula [http://www.mdcalc.com/creatinine-clearance-cockcroft-gault-equation/])
5. Recovery (to baseline or to Grade 1 or less) from prior treatment-related toxicities
6. Ability to swallow capsules
7. Ability to comply with treatment, laboratory monitoring and required clinic visits
8. Able to understand and willing to sign the informed consent form (ICF)

In addition, the following criteria must be met based on the group to be enrolled into:

For subjects in the Phase 1 Single Agent CGX1321 Dose Escalation phase:

1. Pathologically-confirmed, locally advanced or metastatic solid tumors in subjects that have relapsed or are refractory to or are not considered medically suitable to receive standard of care treatment
2. Eastern Cooperative Oncology Group (ECOG) score of 0 - 2
3. Willingness for subjects of reproductive potential to use adequate methods of contraception during and for 3 months after study treatment

For subjects in the Phase 1 Single Agent CGX1321 Dose Expansion phase:

1. Histologically diagnosed advanced GI tumors, such as colorectal adenocarcinoma, gastric adenocarcinoma, pancreatic adenocarcinoma, bile duct carcinoma, hepatocellular carcinoma, esophageal carcinoma in subjects that have relapsed or are refractory to or are not considered medically suitable to receive standard of care treatment. Subjects must have confirmed genetic alterations (e.g., Rspo2 fusion, Rspo3 fusion or predicted loss-of-function mutations in RNF43) upstream in the WNT pathway and no predicted change-of-function alterations in genes (e.g., APC, CTNNB1 and Axin1) downstream in the WNT pathway
2. ECOG score of 0 - 2
3. Willingness for subjects of reproductive potential to use adequate methods of contraception during and for 3 months after study treatment

For subjects in the Phase 1b or Roll-over Cohort CGX1321 in combination with pembrolizumab:

1. Histologically or cytologically confirmed diagnosed advanced colorectal tumors that are mismatch repair-proficient or MSS in subjects that have relapsed or are refractory to or are not considered medically suitable to receive standard of care treatment (for dose escalation) and histologically or cytologically confirmed diagnosed advanced colorectal tumors with confirmed genetic alterations (e.g., Rspo2 fusion, Rspo3 fusion or predicted loss-of-function mutations in RNF43) upstream in the WNT pathway and no predicted change-of-function alterations in genes (e.g., APC, CTNNB1 and Axin1) downstream in the WNT pathway (for dose expansion) Note: Not applicable for subjects entering Roll-over Cohort
2. Previous enrollment into either Phase 1 single agent dose escalation or Phase 1 single agent dose expansion with documented disease progression while on treatment with single agent CGX1321 Note: Not applicable for subjects entering Phase 1b
3. ECOG score of 0 - 1
4. Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile or abstain from heterosexual activity for the course of the study through 120 days after the last dose of pembrolizumab. Subjects of childbearing potential are those who have not been surgically sterilized or have been free from menses for > 1 year.

Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject Female subjects of childbearing potential must have a negative serum pregnancy test within 72 hours prior to receiving the first dose of study treatment Male subjects of childbearing potential must agree to use an adequate method of contraception starting with the first dose of pembrolizumab through 120 days after the last dose of pembrolizumab Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject

For subjects in the Phase 1b Cohort CGX1321 in Combination with Encorafenib + Cetuximab:

1. Histologically diagnosed advanced colorectal tumors (CRC) carrying a BRAF V600E mutation in tumor tissue, (as detected by an FDA-approved test) with confirmed genetic alterations (e.g., Rspo2 fusion, Rspo3 fusion or predicted loss-of-function mutations in RNF43) upstream in the WNT pathway and no predicted change-of-function alterations in genes (e.g., APC, CTNNB1 and Axin) downstream in the WNT pathway
2. Have relapsed or are refractory to or are not considered medically suitable to receive standard of care treatment in the metastatic setting Note: Prior treatment with encorafenib + cetuximab is will be is permitted Exclusion Criteria

All subjects must be excluded from participating in the study if subjects meet any of the following criteria:

1. Prior exposure to a WNT inhibitor. Note: Not applicable for subjects entering Roll-over Cohort
2. Received any of the following within the specified time frame prior to administration of study drug:

   • Previous therapy for malignancy within 21 days, including any investigational agents, chemotherapy, immunotherapy, biological or hormonal therapy Note: Only applicable for subjects in single-agent dose escalation cohorts
3. Major surgery within 4 weeks of first dose of study treatment
4. Radiotherapy within 2 weeks of first dose of study treatment. Note for Phase 1b or Roll-over Cohorts: Subjects must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-CNS disease.
5. Significant GI or variceal bleeding or subdural hematoma within 3 months of first dose of study treatment
6. Known active central nervous system metastases and/or carcinomatous meningitis Note: Subjects with previously treated brain metastases may participate provided they are radiographically stable (without evidence of progression by imaging (using the identical imaging modality for each assessment, either magnetic resonance imaging [MRI] or computed tomography [CT] scan) for at least four weeks prior to the first dose of study treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 14 days prior to the first dose of study treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability
7. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone or equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug
8. Currently receiving medications known to be inhibitors of CYP3A4/5. Subjects currently receiving medications of known inducers of CYP3A4/5 or substrates of CYP2C8/9 and CYP1A2 may be excluded unless determined by the Investigator to be in the best interest of the subject and are approved by the Sponsor
9. Osteoporosis based on a T-score of < -2.5 at the left or right total hip, left or right femoral neck or lumbar spine (L1 - L4) as determined by dual-energy x-ray absorptiometry (DXA) scan
10. Subjects with bone metastases that:

    * Have a prior history of a pathologic fracture
    * Have a lytic lesion requiring an orthopedic intervention or
    * Are not receiving a bisphosphonate (zoledronic acid or denosumab) as per institutional guidelines
11. Current bisphosphonate therapy for symptomatic hypercalcemia
12. History within last 6 months of New York Heart Association Class III or IV heart failure, acute myocardial infarction, angina pectoris, uncontrolled arrhythmia, acute coronary syndromes, stent placement, uncontrolled hypertension
13. Subjects with QTc interval of > 470 msec
14. Known human immunodeficiency virus positive (such patients are at increased risk of lethal infections when treated with potentially marrow-suppressive therapy)
15. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer
16. Active systemic infection requiring IV antibiotics within 2 weeks of the first dose of study treatment
17. History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating Investigator
18. Known psychiatric or substance abuse disorders that would interfere with the subject's ability to cooperate with the requirements of the study.
19. Pregnancy or lactation
20. Has had an allogeneic tissue/solid organ transplant

In addition, subjects must be excluded from participating if they meet any of the following criteria based on the group to be enrolled into:

For subjects in the Phase 1 Single Agent CGX1321 Dose Escalation or Dose Expansion phase:

1. Known active hepatitis A, B or C Note: Subjects who are HBsAg+ and have DNA load < 2000 IU/mL (104 copies/mL) are eligible to participate in the Phase 1 study

For subjects in the Phase 1b or Roll-over Cohort CGX1321 in combination with pembrolizumab:

1. Has a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as HCV RNA [qualitative] is detected) infection.

   Note: No testing for Hepatitis B and Hepatitis C is required unless mandated by local health authority
2. Received transfusion of blood products (including platelets or red blood cells) or administration of colony stimulating factors (including G-CSF, GM-CSF or recombinant erythropoietin) within 4 weeks prior to first dose of study treatment
3. Active autoimmune disease that has required systemic treatment in past 2 years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment
4. History of (non-infectious) pneumonitis that required steroids or current pneumonitis
5. History of interstitial lung disease
6. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of study treatment
7. Received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g., CTLA-4, OX 40, CG137) and was discontinued from that treatment due to a Grade 3 or higher irAE or if the patient has previously participated in Merck MK-3475 clinical studies
8. Has severe (≥ Grade 3) hypersensitivity to any of the excipients of pembrolizumab
9. Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from AEs due to agents administered more than 4 weeks earlier
10. Received a live-virus vaccination within 30 days of planned treatment start. Seasonal flu vaccines that do not contain live virus are permitted

For subjects in the Phase 1b Cohort CGX1321 in Combination with Encorafenib + Cetuximab:

1. Symptomatic brain metastases or leptomeningeal disease
2. History or current evidence of retinal vein occlusion or current risk factors for retinal vein occlusion (e.g., uncontrolled glaucoma or ocular hypertension, history of hyperviscosity or hypercoagulability syndromes)
3. Known history of acute or chronic pancreatitis
4. History of chronic inflammatory bowel disease or Crohn's disease requiring medical intervention (immunomodulatory or immunosuppressive medications or surgery) ≤12 months prior to enrollment
5. Uncontrolled blood pressure despite medical treatment
6. Impaired GI function or disease that may significantly alter the absorption of encorafenib (e.g., ulcerative diseases, uncontrolled vomiting, malabsorption syndrome, small bowel resection with decreased intestinal absorption)
7. History of thromboembolic or cerebrovascular events ≤ 6 months prior to starting study treatment including transient ischemic attacks, cerebrovascular accidents, deep vein thrombosis or pulmonary emboli
8. Concurrent neuromuscular disorder that is associated with the potential of elevated creatinine (phosphor)kinase (CK) (e.g., inflammatory myopathies, muscular dystrophy, amyotrophic lateral sclerosis, spinal muscular atrophy)
9. Active hepatitis B or hepatitis C infection
10. Known history of Gilbert's syndrome
11. Known contraindication to receive Encorafenib or Cetuximab at the planned doses

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2016-02 (Actual); Primary Completion 2023-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events and/or abnormal laboratory values that are related to treatment | 55 months
  safety

SECONDARY OUTCOMES:
CGX1321 area under the curve | 30 Days
  pharmacokinetics
CGX1321 maximum or peak concentration | 30 Days
  pharmacokinetics
CGX1321 minimum or trough concentration | 30 Days
  pharmacokinetics
CGX1321 time to maximum concentration | 30 Days
  pharmacokinetics
CGX1321 half-life | 30 Days
  pharmacokinetics

CONTACTS AND LOCATIONS:
Locations (26):
- United States (25):
  - Memorial Care, Long Beach, California
  - St. Joseph's Santa Rosa, Santa Rosa, California
  - Sarah Cannon Research Institute at HealthONE, Denver, Colorado
  - Hartford Health Care, Hartford, Connecticut
  - Lombardi Comprehensive Cancer Center, Washington D.C., District of Columbia
  - Brooksville, Florida
  - CSNF Cancer Specialists of North Florida (QCCA), Jacksonville, Florida
  - Ocala Oncology, Ocala, Florida
  - University Cancer & Blood Center (QCCA), Athens, Georgia
  - Hawaii Cancer Center, Honolulu, Hawaii
  - Edward H. Kaplan MD and Associates, Skokie, Illinois
  - Goshen Health, Goshen, Indiana
  - Community Health Network, Indianapolis, Indiana
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Nebraska Cancer Specialists (QCCA), Omaha, Nebraska
  - Summit Medical Group, Florham Park, New Jersey
  - Duke Cancer Center, Duke University Medical Center, Durham, North Carolina
  - Gettysburg Cancer Center, Gettysburg, Pennsylvania
  - Sanford Health, Sioux Falls, South Dakota
  - Baptist Cancer Center, Memphis, Tennessee
  - START (South Texas Accelerated Research Therapeutics, LLC), San Antonio, Texas
  - Northwest Medical Specialists (QCCA), Tacoma, Washington
  - University of Wisconsin Carbone Cancer Center, Madison, Wisconsin
- Taipei Medical University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No